CLINICAL TRIAL: NCT02400658
Title: A Prospective Single-Arm Phase II Study To Investigate The Efficacy Of Single-Fraction Intraoperative Radiation Treatment Using A Multi-Lumen Balloon Applicator And In-Room CT Imaging For The Treatment Of Early-Stage Breast Cancer
Brief Title: Efficacy of IORT With CT-Guided HDR Brachytherapy for Treatment of Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shayna Showalter, MD (Other)
Responsible Party: Sponsor-Investigator, Shayna Showalter, MD, Assistant Professor of Medicine, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18004; IORT2 (Other: University of Virginia)
Record Dates: First submitted 2015-03-12; First posted 2015-03-27 (Estimated); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; early-stage; IORT; brachytherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative; Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IORT with CT-Guided HDR Brachytherapy (Experimental): Patients will receive IORT with CT-guided HDR brachytherapy at the time of breast surgery.
  Interventions: Device: IORT with CT-Guided HDR Brachytherapy

INTERVENTIONS:
Device: IORT with CT-Guided HDR Brachytherapy — This therapy targets the cancer cells directly, reducing the volume of breast tissue exposed to the radiation and the risks involved with the radiation. CT imaging will be used via a multichannel/multi-dwell balloon catheter to better sculpt the cancer away from the heart, skin, and ribs.
  Other Names: Surgery; Breast Lumpectomy

SUMMARY:
The purpose of this study is to evaluate an investigational way to provide radiation therapy to treat early-stage breast cancer at the time of surgery.

DETAILED DESCRIPTION:
This is a prospective single-arm phase II study designed to study the efficacy of high dose rate (HDR) brachytherapy with CT-imaging, single-fraction intraoperative radiation therapy (IORT). The study will accrue patients with early-stage breast cancer who will be treated with breast-conserving surgery (BCS). The main clinical eligibility criterion is based on suitability for accelerated partial breast irradiation. Patients may be eligible prior to receiving BCS or within 30 days of receiving BCS. Eligible patients that will undergo BCS will receive surgery according to the standard clinical practice in the Brachytherapy Suite in the Emily Couric Clinical Cancer Center. Patients that have already undergone BCS must meet all other eligibility criteria and are able to be treated with IORT within 30 days of their breast surgery. Eligible subjects will undergo a lumpectomy or re-excision lumpectomy according the standard clinical practice. Immediately following lumpectomy, the breast HDR brachytherapy applicator will be placed and CT imaging will be performed for treatment planning. After HDR brachytherapy is delivered, the applicator will be removed, and the breast surgeon will complete the skin closure. Although the ultimate goal of the study is to determine 5-year ipsilateral breast tumor recurrence (IBTR), all efforts will be made to follow the patients until death.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has elected breast conserving surgery or whole breast irradiation treatment for early-stage breast cancer.
2. Tumor size must be less than or equal to 3 cm.
3. Patient is 45 years of age or older.

Exclusion Criteria:

1. Male patients.
2. Pregnant patients.
3. Breast cancer that involves the skin or chest wall.
4. History of ipsilateral breast cancer.
5. Multicentric breast cancer in the ipsilateral breast.
6. Known BRCA gene mutation.
7. Patient with nodal disease.
8. Patient is undergoing initial medical treatment (hormone or chemotherapy) to reduce tumor size.
9. Patient with breast implants (does not include patients having implants AFTER intra-operative radiotherapy).

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2015-03; Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Local Breast Tumor Recurrence | Up to 60 Months After Treatment

SECONDARY OUTCOMES:
Rate of Ipsilateral Breast Tumor (Not Local) Recurrence | Up to 60 Months After Treatment
Rate of Distant Recurrence of Breast Cancer | Up to 60 Months After Treatment
Cancer Specific-Survival and Overall Survival Response Rate | Minimum of 60 Months After Treatment
Changes in Reported Patient and Physician Cosmetic Descriptions | Up to 60 Months After Treatment
Comparison of Pre-and Post Pathology Stratum | Up to 60 Months After Treatment
Changes in Patient-Reported Quality of Life | Up to 60 Months After Treatment
Number of Participants with Adverse Events | 24 Months After Treatment
  Safety and toxicity of treatment will be determined with the Common Toxicity Criteria for Adverse Effects.
Changes of Radiographic Breast Appearance | Up to 60 Months After Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shayna Showalter, Principal Investigator — University of Virginia
Locations (3):
- United States (3):
  - Hackensack Meridian Health - John Theurer Cancer Center, Hackensack, New Jersey
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Turkheimer LM, Petroni GR, Berger AC, Schroen AT, Brenin DR, Lazar M, Libby B, Janowski EM, Showalter TN, Showalter SL. Novel Form of Breast Intraoperative Radiation Therapy with CT-Guided High-Dose-Rate Brachytherapy: Interim Results of a Prospective Phase-II Clinical Trial. J Am Coll Surg. 2024 Jan 1;238(1):10-20. doi: 10.1097/XCS.0000000000000869. Epub 2023 Oct 23. PMID 37870228
- [Derived] Meneveau MO, Petroni GR, Varhegyi NE, Hulse JC, Schroen AT, Brenin DR, Janowski EM, Berger AC, Lazar MA, Simone NL, Showalter TN, Showalter SL. Toxicity and cosmetic outcomes after treatment with a novel form of breast IORT. Brachytherapy. 2020 Sep-Oct;19(5):679-684. doi: 10.1016/j.brachy.2020.05.002. Epub 2020 Jun 20. PMID 32571746